CLINICAL TRIAL: NCT06637241
Title: Compare the Effectiveness of Injury Prevention Between Risk Stratification Care and Usual Care in Taiwan Adolescent Baseball Players: a Cluster Randomized Controlled Trial.
Brief Title: Risk Stratification Care for Injury Prevention in Taiwan Adolescent Baseball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG8P0161
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Adolescent Baseball Players
Keywords: Throwing arm injury; Stratified care for injury risk; Long term follow up; Health-related quality of care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Schools assigned to the usual care management group will receive a visit from one of the co-principal investigators, who will explain the project to the coaches and athletic trainers but request that they do not change their existing training plans or care practices. However, medical consultation or referral contact information will be provided if needed.
- Risk stratification care (Experimental): All baseball players at schools assigned to the injury risk-stratified care group will be categorized into high-risk, medium-risk, and low-risk groups. Baseball players in the high-risk group will receive not only sports protection education but will also be referred to a physician for further care. The sports protective education is taught by a sports injury prevention specialist from the Sports Injury Prevention System for Student Athletes of the Sports Administration. This education includes a prevention program known as the Modified Yokohama Baseball-9 (mYKB-9), which has been clinically validated to effectively reduce shoulder and elbow joint injuries in adolescent baseball players by nearly half. The program consists of nine exercises, including five stretches, two thoracic mobility exercises, and two lower limb balance exercises.
  Interventions: Behavioral: Risk stratification care

INTERVENTIONS:
Behavioral: Risk stratification care — In this group, Taiwanese adolescent baseball players are categorized into high-risk, medium-risk, and low-risk groups based on injury risk from a previous study. High-risk players receive sports protection education and physician referrals for shoulder and elbow assessments, with further imaging if necessary. Common issues like Little League shoulder and elbow are managed with conservative treatments. The sports protection education includes the Modified Yokohama Baseball-9 (mYKB-9), a program that significantly reduces injuries with exercises targeting shoulder and elbow health. Medium-risk players receive mYKB-9 education only, while low-risk players are observed without changes to their training methods.
  Arms: Risk stratification care

SUMMARY:
Due to frequent practices and competitions, Taiwanese adolescent baseball players gradually accumulate fatigue, leading to injuries in their throwing arms. Previous research on baseball has primarily focused on the epidemiology of sports injuries, biomechanical analysis of throwing motions, and the effectiveness of injury prevention interventions. Based on our previous research on the quality of life of Taiwanese adolescent baseball players, we have gained a general understanding of the impact of throwing arm injuries on these athletes. This study aims to stratify the injury risks of these baseball players based on past research and provide corresponding care guidelines according to different risk levels. We will compare this care model with standard care through a cluster randomized controlled trial, aiming to verify that this model is effective, efficient, and more clinically applicable than previous injury prevention interventions. Ultimately, we hope to promote this care model across all youth baseball teams in Taiwan.

DETAILED DESCRIPTION:
Baseball involves repetitive throwing motions that place considerable stress on the shoulder and elbow, leading to throwing arm injuries. Previous studies have shown that baseball players are at a higher risk of upper limb injuries compared to the general population, particularly pitchers. In Major League Baseball (MLB) in the United States, more than half of the injuries are to the upper limbs, and 48.4% of these are caused by throwing motions. Since throwing is a crucial part of baseball, injuries to the throwing arm can result in significant disability, both in sports and non-sports contexts. These disabilities not only affect the performance of baseball players but also have broader implications, including psychological and social impacts.

Recently, the importance of patient-reported outcomes (PRO) in clinical research has been increasingly recognized. In the past, clinical assessments focused primarily on physician evaluations of physical examinations and diagnostic test results. However, these measures may not accurately reflect patients' actual experiences. PROs can help physicians assess patients' health-related quality of life (HRQOL). This concept has also started to gain traction in the field of sports medicine.

Taiwanese adolescent baseball players face varying degrees of injury risk based on their defensive positions. In addition, measuring HRQOL may help identify injury risks that cannot be determined solely by their defensive positions. For high-risk baseball players, early referral to a physician for further examination and treatment can greatly aid in preventing injuries or facilitating recovery and return to the field after an injury. To identify high-risk individuals among a group of baseball players, our research team has collaborated with several junior high and high school baseball teams in Kaohsiung (including seven junior high schools and one high school).

ELIGIBILITY:
Inclusion Criteria:

1. All youths who are members of their school's baseball team and are willing to participate in the study with parental consent.
2. Agree to participate in the trial and complete the participant consent form.

Exclusion Criteria:

(1) A history of significant musculoskeletal or neurological injuries (or functional abnormalities).

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Functional Arm Scale for Throwers (FAST) | From enrollment to the end of study at 12 months.
  This study strives to observe changes in the quality of life among Taiwanese adolescent baseball players over the course of a year. To achieve this, the questionnaire will be administered multiple times, with visits to the schools for measurements once per season (every 3 months). The primary measurement tool will be the Chinese version of the FAST scale, which has been validated in preliminary research.

SECONDARY OUTCOMES:
Injury | From enrollment to the end of the study at 12 months
  Each season, during school visits, the study will examine baseball players in the team who have experienced throwing arm injuries. Coaches will be asked to identify players who have had injuries in the past three months and refer them to the visiting physician for assessment. If physical examination and ultrasound screening confirm abnormalities in the shoulder (such as rotator cuff tendinitis or tears, shoulder labral injuries, etc.) or elbow (such as medial epicondylitis, ulnar collateral ligament injuries, osteochondritis dissecans, etc.), the player will be classified as injured. Injury data will be categorized as follows: injury occurrence (dichotomous data), number of injuries (count data), and severity (ordinal data). The number of injuries will be determined by asking players how many times they have experienced throwing arm injuries in the past three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Secondary analysis might be performed after the primary study, so IPD will not be shared immediately after finishing the study.